CLINICAL TRIAL: NCT03954977
Title: Point of Care Ultrasound for PICC Line Monitoring Study
Acronym: PUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Patrick Motz, Neonatal Perinatal Fellow, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0503
Record Dates: First submitted 2019-04-28; First posted 2019-05-17 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Peripherally Inserted Central Catheters
Keywords: PICC line; Neonate

STUDY DESIGN:
Intervention Model Description: A prospective comparative study evaluating chest x-ray determination of PICC line tip location and POC ultrasound PICC line tip location. NICU patient's with PICC lines will be enrolled and blinded ultrasound operators will scan the neonate to find the PICC tip location. This will be compared to the location on the patient's chest x-ray. This process will be repeated each time the patient has a chest x-ray.
Masking Description: Investigator is blinded to xray result before doing ultrasound
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ultrasound vs Radiograph (Experimental): NICU patient's with PICC lines will be enrolled and blinded ultrasound operators will scan the neonate to find the PICC tip location. This will be compared to the location on the patient's chest x-ray. This process will be repeated each time the patient has a chest x-ray.
  Interventions: Diagnostic Test: PICC line ultrasound

INTERVENTIONS:
Diagnostic Test: PICC line ultrasound — NICU patient's with PICC lines will be enrolled and blinded ultrasound operators will scan the neonate to find the PICC tip location. This will be compared to the location on the patient's chest x-ray. This process will be repeated each time the patient has a chest x-ray.

SUMMARY:
A prospective comparative study evaluating chest x-ray determination of PICC line tip location and POC ultrasound PICC line tip location. NICU patient's with PICC lines will be enrolled and blinded ultrasound operators will scan the neonate to find the PICC tip location. This will be compared to the location on the patient's chest x-ray. This process will be repeated each time the patient has a chest x-ray.

DETAILED DESCRIPTION:
Point of care (POC) ultrasound has become an invaluable tool for critically ill children. Several studies have been completed detailing its use for central line access and determining the location of the tip of umbilical venous lines. There are no current studies on monitoring PICC line tip placement using POC ultrasound. There have been studies showing ultrasound can be used to locate PICC line tip location, but none for monitoring. A previous study found that the sensitivity and specificity of US in identifying the location of PICC line tip were 86% and 75% respectively.

Review of the literature notes that Costa et al also found a high rate of PICC line complications. Costa et al and the investigators local experience also highlight the rare but potentially fatal complication of pericardial effusion from PICC lines that are too deep in the heart. One way the investigators could improve the safety of neonatal PICC lines is monitor them more closely. Current standard of care is to monitor PICC line tips on chest x-ray. Unfortunately, there is strong evidence that chest x-ray does not accurately identify the PICC line tip location. Another way would be to use POC ultrasound. A literature review on POC ultrasound to determine the location of a PICC line tip revealed that no such study has been done. Several studies have been completed demonstrating POC ultrasound both improved success rate and time to confirmation of placement of PICC lines.3 Pulickal et al published data on teaching pediatric residents to do point of care ultrasound to determine the location of the UVC tip. The investigators in that study found the residents were not only better at determining the correct location than chest x-ray, but the procedure was well tolerated. The investigators for this study feel further evaluation of POC ultrasound for PICC line tip monitoring to determine feasibility and accuracy is needed.

Eligible patients will be identified by the NICU care team. Participants will then be consented for the study by the study team. Trained Neonatology Fellows/Attendings will perform POC ultrasound to identify and document the PICC tip location and will be blinded to the PICC line tip location on x-ray. Ultrasounds will only be performed during patient's care times and be limited to 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* NICU patient at Seattle Childrens Hospital or University of Washington
* Patient has a PICC line in place

Exclusion Criteria:

* vertebral anomalies
* anomalies of venous anatomy
* tracheal anomalies.

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
PICC line tip is located by the ultrasound operator | 6 months
  PICC line identified under ultrasound

SECONDARY OUTCOMES:
PICC line location on ultrasound agrees with radiograph | 6 months
  PICC line localization on ultrasound is the same as the localization of the PICC line on radiograph

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Seattle Childrens Hospital, Seattle, Washington
  - University Of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No